CLINICAL TRIAL: NCT01059968
Title: The Role of Low Energy Availability and the H-P-A Axis, Menstrual Irregularity, and Low Bone Mass
Brief Title: Low Energy Availability, Menstrual Irregularity, and Low Bone Mass
Status: Completed | Type: Observational
Sponsor: USDA, Western Human Nutrition Research Center (U.S. Federal Agency)
Collaborators: San Diego State University (Other)
Responsible Party: Marta Van Loan, USDA, ARS, Western Human Nutrition Research Center
Other Study IDs: 200816305-1
Record Dates: First submitted 2009-12-28; First posted 2010-02-01 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2011-06

CONDITIONS: Bone Density; Energy Availability
Keywords: bone density; energy availability; menstrual status; female; adolescent

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- adolescent female endurance athletes: High school female cross country runners in San Diego.

SUMMARY:
This study examines the role of energy availability on menstrual function and bone mass in female adolescent endurance athletes. Specific evaluations include dietary intake, exercise energy expenditure, training schedules, menstrual function and bone density.

DETAILED DESCRIPTION:
The purpose of this project is to examine the relationships among low energy availability, H-P-A axis, menstrual function and bone density and bone turnover in high school female cross country runners. Our objectives are to: 1)determine energy intake, exercise energy expenditure, and fat-free mass to examine energy availability; 2)in a subset of runners, using double labelled water, estimate total energy expenditure and indirect calorimetry to estimate resting metabolic rate; 3)assess the relationship between energy availability, hormones that regulate bone turnover, markers of bone formation and resorption and bone mineral content and density; 4)identify the relationship between energy availability, hormones that regulate menstrual function and current menstrual status; and 5)determine the energy intake and energy expenditure variables exhibiting the strongest associations with energy availability.

ELIGIBILITY:
Inclusion Criteria:

* high school female cross country runners
* ages 15-17 years
* 1-5 years experience as cross country runner
* 25 miles or more/week training

Exclusion Criteria:

* medications known to affect bone metabolism
* pregnancy

Ages: 15 Years to 17 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Study Population: adolescent female cross country runners
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2008-09; Primary Completion 2008-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Bone density | 3 months

SECONDARY OUTCOMES:
Energy availability | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Marta D Van Loan, Ph.D., Study Chair — USDA, ARS, Western Human Nutrition Research Center
Locations (1):
- Marta Van Loan, Davis, California, United States

REFERENCES:
- [Derived] Wood KL, Barrack MT, Gray VB, Cotter JA, Van Loan MD, Rauh MJ, McGowan R, Nichols JF. Cognitive dietary restraint score is associated with lower energy, carbohydrate, fat, and grain intake among female adolescent endurance runners. Eat Behav. 2021 Jan;40:101460. doi: 10.1016/j.eatbeh.2020.101460. Epub 2020 Nov 25. PMID 33307469
- [Derived] Barrack MT, Van Loan MD, Rauh MJ, Nichols JF. Physiologic and behavioral indicators of energy deficiency in female adolescent runners with elevated bone turnover. Am J Clin Nutr. 2010 Sep;92(3):652-9. doi: 10.3945/ajcn.2009.28926. Epub 2010 Jul 7. PMID 20610635